CLINICAL TRIAL: NCT01552226
Title: Prospective Randomized Clinical Trial to Compare Continuous Preperitoneal Analgesia to Continuous Epidural Analgesia for Pain Control After Colon and Rectal Surgery
Brief Title: Compare Preperitoneal Analgesia to Epidural Analgesia for Pain Control After Colon and Rectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCNM 114
Record Dates: First submitted 2012-02-28; First posted 2012-03-13 (Estimated); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer; Rectal Cancer; Colonic Diverticulosis
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Diverticulosis, Colonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Preperitoneal Analgesia (CPA) (Active Comparator): Continuous Preperitoneal Analgesia for pain management
  Interventions: Device: Continuous Preperitoneal Analgesia
- Continuous Epidural Analgesia (CEA) (Active Comparator): Continuous Epidural Analgesia for pain management
  Interventions: Device: Continuous Epidural Analgesia

INTERVENTIONS:
Device: Continuous Preperitoneal Analgesia — Preperitoneal catheter placed at the completion of surgery in the standard fashion.
  Other Names: On-Q Silver Soaker(tm)
  Arms: Continuous Preperitoneal Analgesia (CPA)
Device: Continuous Epidural Analgesia — Epidural catheter placed prior to the operation in the standard fashion.
  Arms: Continuous Epidural Analgesia (CEA)

SUMMARY:
This is a prospective randomized study of 114 patients. The purpose of this study is to compare the efficacy of two standard methods of analgesia for pain control in patients undergoing elective colon and rectal surgery, as measured by the Numeric Pain Scale (NPS) and by the need for supplemental narcotic analgesics. This study is designed to determine if postoperative pain control by local analgesics delivered through preperitoneally placed ON-Q Silver Soaker™ catheters (CPA) is equivalent to continuous epidural analgesia (CEA).

DETAILED DESCRIPTION:
Background Perioperative analgesia is a vital part of the management of patients undergoing colon and rectal surgery, affecting well being and length of hospital stay. Neuraxial anesthetics infused through epidural or spinal catheters have become commonplace pain management agents for patients. These techniques, however, are labor-intensive and expensive. Alternatively, local analgesics may be administered directly to the surgical wound via silver catheters.

Aim Two standard methods of analgesia for pain control for colon and rectal surgery will be evaluated systematically to determine if these two approaches are equivalent in terms of patient pain scores and supplemental narcotic use.

Study Design This is a prospective randomized study of 114 participants undergoing elective colon and rectal surgery at an independent academic medical center. The primary outcomes are post-operative pain control and supplemental narcotic usage.

Other variables of interest

* Surgical site infections
* The post-operative time to return of bowel function
* The hospital expenses/cost differences
* Quality of life measured with the Short Form (SF)- 36 questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age > = 18 years
* Scheduled for elective colon or rectal surgery
* Surgical procedure either through open laparotomy or via minimal invasive approach (laparoscopic)
* Able to provide informed consent
* Able to complete patient questionnaire

Exclusion Criteria:

* Documented allergic reaction to morphine, hydromorphone, lidocaine, bupivicaine and/or fentanyl
* Contra-indication to placement of epidural catheter (spinal stenosis, spinal fusion, etc)
* Urgent surgery precluding epidural catheter placement
* Systemic Infection contraindicating epidural catheter placement
* Unwillingness to participate in follow up assessments
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cleary, MD, Principal Investigator — Trinity Health Michigan
Locations (1):
- Saint Joseph Mercy Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- See also: American Society of Colon and Rectal Surgeons — http://www.fascrs.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Started | 50 | 48
Completed | 46 | 44
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA) | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.2) | 60.8 (12.6) | 60.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 28 | 23 | 51
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is measured by a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
  kg/m^2 | 29.1 (6.6) | 29.6 (5.9) | 29.35 (6.25)
Tobacco Use [Count of Participants; unit: Participants] | 8 | 4 | 12
Narcotics use [Count of Participants; unit: Participants] | 4 | 2 | 6
Diabetes [Count of Participants; unit: Participants] | 4 | 3 | 7
Blood thinners [Count of Participants; unit: Participants] | 3 | 3 | 6
Primary diagnosis [Count of Participants; unit: Participants]
  Malignancy | 21 | 24 | 45
  Diverticulitis | 19 | 13 | 32
  Irritable Bowel Disease | 2 | 3 | 5
  Other | 4 | 4 | 8
Surgical approach [Count of Participants; unit: Participants]
  Open | 8 | 6 | 14
  Laparoscopic | 3 | 2 | 5
  Robotic | 35 | 36 | 71
Procedure Type [Count of Participants; unit: Participants]
  Partial Colectomy | 33 | 35 | 68
  Lower Pelvic Anastomosis | 13 | 9 | 22
Wound class II, clean contaminated [Count of Participants; unit: Participants] — Patients are "graded" based on standardized definitions of wound classes and are assigned these grades during debriefing after skin closure. This grade is then documented in the patient record.
  Class II/Clean-Contaminated: An operative wound in which the respiratory, alimentary, genital, or urinary tracts are entered under controlled conditions and without unusual contamination. Specifically, operations involving the biliary tract, appendix, vagina, and oropharynx are included in this category, provided no evidence of infection or major break in a sterile technique is encountered.
  Participants | 45 | 43 | 88
Preoperative Short Form Health Survey (SF-36 subscale) [Mean (Standard Deviation); unit: units on a scale] — Preoperative Short Form Health Survey refers to a set of questions from the SF-36 that a patient completes before a surgical procedure, with an overall aggregate scale and eight subscales. The subscales assess aspects of their health status, including physical functioning, bodily pain, role limitations due to physical health, social functioning, mental health, vitality, and general health perceptions, allowing healthcare providers to understand the patient's baseline health condition before surgery. Each subscale is scored on a scale from 0 to 100, with higher scores indicating better health. Population: The numbers are different due to the difference in number of respondents on some of the sub scales.
  units on a scale
    Aggregate score: number analyzed (Participants) | 44 | 42 | 86
    Aggregate score | 74.7 (14.6) | 67.0 (17.9) | 70.8 (16.2)
    Physical functioning: number analyzed (Participants) | 44 | 41 | 85
    Physical functioning | 83.3 (21.4) | 73.3 (26.0) | 78.3 (23.7)
    Role limitations: physical health: number analyzed (Participants) | 8 | 10 | 18
    Role limitations: physical health | 65.6 (48.1) | 55.0 (49.7) | 60.3 (48.9)
    Role limitations: emotional problems: number analyzed (Participants) | 4 | 5 | 9
    Role limitations: emotional problems | 75.0 (50.0) | 60.0 (54.8) | 67.5 (52.4)
    Energy: number analyzed (Participants) | 42 | 41 | 83
    Energy | 61.8 (17.0) | 55.3 (18.8) | 58.5 (17.9)
    Emotional: number analyzed (Participants) | 42 | 41 | 83
    Emotional | 69.5 (13.2) | 64.6 (19.0) | 67.0 (16.1)
    Social: number analyzed (Participants) | 44 | 42 | 86
    Social | 84.1 (23.9) | 75.0 (27.3) | 79.5 (25.6)
    Pain: number analyzed (Participants) | 43 | 42 | 85
    Pain | 76.4 (27.5) | 74.1 (23.4) | 75.2 (25.4)
    General health: number analyzed (Participants) | 44 | 42 | 86
    General health | 70.7 (19.1) | 65.4 (21.0) | 68.0 (20.0)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Numerical Pain Score-Day 0
Description: Measured by the patient using the numerical pain scale (NPS). NPS is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Time Frame: Post-operative day 0
Population: The Overall Number of Participants Analyzed is not consistent with the numbers provided in the Participant Flow module. This discrepancy is due to the difference in the number of respondents on this scale for this timeframe.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 45 | 44
units on a scale | 3.9 (2.0) | 2.6 (1.7)

2. Primary Outcome: Postoperative Numerical Pain Score-Day 1
Description: as for outcome 1
Time Frame: Post-operative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 46 | 44
units on a scale | 3.2 (1.8) | 2.6 (1.9)

3. Primary Outcome: Postoperative Numerical Pain Score-Day 2
Description: as for outcome 1
Time Frame: Post-operative day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 45 | 43
units on a scale | 2.6 (1.7) | 2.1 (1.7)

4. Primary Outcome: Postoperative Numerical Pain Score-Day 3
Description: as for outcome 1
Time Frame: Post-operative day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 37 | 39
units on a scale | 2.9 (1.9) | 2.7 (1.9)

5. Primary Outcome: Postoperative Numerical Pain Score-Day 4
Description: as for outcome 1
Time Frame: Post-operative day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 26 | 26
units on a scale | 3.1 (2.1) | 2.7 (1.8)

6. Primary Outcome: Postoperative Numerical Pain Score (NPS)- Post-Anaesthesia Care Unit (PACU)
Description: Postoperative NPS is a pain screening tool, commonly used to assess the pain severity a patient experiences after surgery, where "0" indicates no pain and "10" represents the worst pain imaginable".
Time Frame: After surgery in the post-anesthesia care unit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 44 | 41
units on a scale | 3.5 (2.8) | 2.3 (2.5)

7. Secondary Outcome: Patient Use of Supplemental Narcotic Analgesia Day 1
Description: Patient use of supplemental narcotic analgesia day 1 measured in morphine equivalents.
Time Frame: Post-operative day 1
Population: "The Overall Number of Participants Analyzed" is not consistent with the numbers provided in the Participant Flow module due to the difference in the number of respondents on the scale.
Measure: Mean (Full Range); unit: Morphine equivalents
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 45 | 44
Morphine equivalents | 29 [20.1 to 41.8] | 23 [14.4 to 36.4]

8. Secondary Outcome: Patient Use of Supplemental Narcotic Analgesia Day 2
Description: Patient use of supplemental narcotic analgesia day 2 measured in morphine equivalents.
Time Frame: Post-operative day 2
Population: as for outcome 1
Measure: Mean (Full Range); unit: morphine equivalents
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 43 | 43
morphine equivalents | 22.4 [14.2 to 35.1] | 21.2 [13.9 to 32.0]

9. Secondary Outcome: Patient Use of Supplemental Narcotic Analgesia Day 3
Description: Patient use of supplemental narcotic analgesia on day 3, measured in morphine equivalents.
Time Frame: Post-operative day 3
Population: as for outcome 1
Measure: Mean (Full Range); unit: morphine equivalents
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 34 | 37
morphine equivalents | 17.4 [10.4 to 28.6] | 16.0 [10.7 to 23.7]

10. Secondary Outcome: Patient Use of Supplemental Narcotic Analgesia Day 4
Description: Patient use of supplemental narcotic analgesia day 4 measured in morphine equivalents.
Time Frame: Post-operative day 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: morphine equivalents
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 29 | 29
morphine equivalents | 6.9 [3.7 to 12.3] | 9.2 [5.1 to 15.9]

11. Secondary Outcome: Patient Use of Supplemental Narcotic Analgesia Day 0
Description: Patient use of supplemental narcotic analgesia day 0 measured in morphine equivalents.
Time Frame: Post-operative day 0
Population: as for outcome 1
Measure: Mean (Full Range); unit: morphine equivalents
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Number analyzed (Participants) | 45 | 44
morphine equivalents | 20.5 [14.2 to 29.5] | 11.0 [7.1 to 16.6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Continuous Preperitoneal Analgesia (CPA) | Continuous Epidural Analgesia (CEA)
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 0/50 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No